CLINICAL TRIAL: NCT06588439
Title: Cognitive-motor Training on Brain Activity, Cognitive Function, and Walking Ability in People With Parkinson Disease
Brief Title: Cognitive-motor Training in Parkinson Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU113006AF2
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Cognitive-motor training; Executive function; Gait; Electroencephalography
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-motor training group (Experimental): Participants receive 16 sessions of cognitive-motor training.
  Interventions: Other: Cognitive-motor training
- Control group (Active Comparator): Participants receive 16 sessions of conventional physiotherapy.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Cognitive-motor training — Cognitive-motor training is that cognitive tasks incorporated into motor tasks.
  Arms: Cognitive-motor training group
Other: Conventional physiotherapy — Conventional physiotherapy includes stretching, ROM exercise, strengthening exercise, and eye-hand coordination.
  Arms: Control group

SUMMARY:
Literature reviews showed the cognitive-motor training that combines cognitive tasks may enhance cognitive functions more effectively than individual interventions. Stepping-based cognitive-motor training has been shown to improve cognitive functions, balance, and gait performance in older adults. However, there is insufficient research evidence on the impact and correlation of this training mode on the walking ability, executive functions, and brain activity changes in people with PD. Therefore, this study is designed to investigate the effects of stepping-based cognitive-motor training on the walking ability, executive functions, and brain activity in people with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of idiopathic Parkinson disease
* Stable dopaminergic medicine ≥ 2 weeks
* Able to walk 10 meters without aid
* Mini-Mental Status Examination ≥ 24 points
* No uncorrected visual or auditory disorders
* Education at least junior high school
* No other disease may affect balance

Exclusion Criteria:

* Other medical diagnoses of neurological, musculoskeletal, or cardiopulmonary disorders
* History of brain surgery (e.g. deep brain stimulation)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Gait variability | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Using GAITRite system to measure the coefficient of variation (CV). The mean and standard deviation will be used to calculate the coefficient of variation (CV). CV = standard deviation / mean * 100%
Gait speed | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Using GAITRite system to measure gait speed
Step length | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Using GAITRite system to measure step length
Step width | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Using GAITRite system to measure step width
Single support time | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Using GAITRite system to measure single support time
Double support time | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Using GAITRite system to measure double support time
Frontal Assessment Battery | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  The score ranged from 0 to 18. Higher scores show better executive function.
Stroop color and word test | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Record numbers of corrected color words which the subject responds within 45 sec.
Digit span test | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Digit span test contain forward and backward part. Scores of forward digit span ranges from 0 to 16. Score of backward digit span ranges from 0 to 14. Higher scores indicate better executive function.
Event-related potential - N2 | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Measure event-related potential through electroencephalography under single-task and dual-task paradigm.
Event-related potential - P300 | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Measure event-related potential through electroencephalography under single-task and dual-task paradigm.
Go/Nogo test | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Behavioral test during measuring electroencephalography.
Trail making test | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Trail making test contain part A and part B. Faster completing the test indicates better executive function.

SECONDARY OUTCOMES:
Mini-Balance Evaluation Systems Test | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Mini-Balance Evaluation Systems Test scores range from 0 to 28. Higher scores indicate better balance ability.
Montreal Cognitive Assessment | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Montreal Cognitive Assessment ranges from 0 to 30. Higher scores reflect better cognitive performances.
Timed up and go test | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Record time of performing timed up and go test
Parkinson Disease Questionnaire | Before and after 8 weeks of intervention, as well as 4 weeks after intervention
  Parkinson Disease Questionnaire assess quality of life in people with Parkinson disease. Lower scores reflect higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan